CLINICAL TRIAL: NCT02981888
Title: Fecal Bile Acids, Fecal Short Chain Fatty Acids and the Intestinal Microbiota in Patients With Irritable Bowel Syndrome and Control Volunteers
Brief Title: Fecal Metabolome and the Intestinal Microbiota in Irritable Bowel Syndrome
Acronym: IBS
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Huiping Xu, Associate Professor, Indiana University
Other Study IDs: 1606244063
Record Dates: First submitted 2016-10-31; First posted 2016-12-05 (Estimated); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: IBS
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- IBS-C: all patients with IBS -C will undergo an abdominal x-ray for assessment of colonic transit
  Interventions: Radiation: X-Ray
- IBS-D: all patients with IBS-D will undergo an abdominal x-ray for assessment of colonic transit
  Interventions: Radiation: X-Ray
- heathy control: all healthy controls will undergo an abdominal x-ray for assessment of colonic transit
  Interventions: Radiation: X-Ray

INTERVENTIONS:
Radiation: X-Ray — X-ray of the abdomen will be performed to assess colonic transit

SUMMARY:
The purpose of this study is to find out the relationship between the bile acids, fatty acids (fatty acids are part of the diet) and bacteria that are present in the intestines.

DETAILED DESCRIPTION:
There is emerging evidence that alterations in bile acids and SCFA associated with IBS could be associated with changes in the gut microbiota. In addition to modulating levels of intraluminal organic acids, it has been hypothesized that gut microbiota may alter local immune responses, modulate visceral pain responses, and impair gut barrier function.

Our overall goal is to investigate the relationship between fecal bile acids, SCFA and the gut microbiota in IBS. Results of this pilot study could reveal insights into the interplay of the gut microbiota and small molecule mediators of IBS to suggest targeted clinical strategies for improved diagnosis and management of this important syndrome.

AIM 1: Test the hypothesis that fecal organic acids (SFCA and bile acids) and fecal microbiota play an important role in IBS.

AIM 2: Test the hypothesis that there is association between colonic transit and fecal microbiota in IBS

ELIGIBILITY:
Inclusion Criteria:

* Patients with IBS, ages 18-65 fulfilling Rome IV criteria and asymptomatic controls with no prior history of GI disease or symptoms.
* Participants should be on a stable and consistent diet regimen and should not be following an extreme diet intervention such as gluten-free or a low FODMAP diet at the time of study participation.

Exclusion Criteria:

* Participants with microscopic/lymphocytic/collagenous colitis, inflammatory bowel disease, celiac disease, visceral cancer, chronic infectious disease, immunodeficiency, uncontrolled thyroid disease, history of liver disease or history of elevated AST/ALT > 2.0x the upper limit of normal
* Prior radiation therapy of the abdomen or abdominal surgeries with the exception of appendectomy or cholecystectomy > 6 months prior to study initiation
* Ingestion of any prescription, over the counter, or herbal medications which can affect GI transit or study interpretation (e.g. opioids, narcotics, anticholinergics, norepinephrine reuptake inhibitors, nonsteroidal anti-inflammatory drugs, COX-2 inhibitors, bile acid sequestrants) within 6 months of study initiation for asymptomatic volunteers or within 2 days before study initiation for IBS patients
* Any females who are pregnant or trying to become pregnant or breast-feeding
* Antibiotic usage within 3 months prior to study participation
* Prebiotic or probiotic usage within the 2 weeks prior to study initiation
* Use of tobacco products within the past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target study population will be patients with IBS (both diarrhea- and constipation-predominant) and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Total and individual fecal bile acid excretion | two days
  Stool samples will be collected over 2 days for measurement of fecal bile acids (µmol/48h) by high performance liquid chromatography-mass spectometry
Total fecal excretion of short chain fatty acids | two days
  Stool samples will be collected for measurement of measurement of short chain fatty acids (µg/mg) by liquid chromatography-mass spectrometry
Fecal microbial population and community from stool collection | two days
  Stool samples will be be collected from participants for nucleic acid extraction, 16S allele PCR and sequencing to measure microbial communities and profiles of specimens

SECONDARY OUTCOMES:
Fecal excretion of individual short chain fatty acids | two days
  Stool samples will be collected for measurement of measurement of short chain fatty acids (µg/mg) by liquid chromatography-mass spectrometry
Stool characteristics | 14 days
  Stool characteristics will be measured using a 14 day bowel diary

OTHER OUTCOMES:
Overall and segmental colon transit | 7 days
  Colonic transit time will be measured in days using radiopaque markers

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Shin, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Waseem MR, Shin A, Siwiec R, James-Stevenson T, Bohm M, Rogers N, Wo J, Waseem L, Gupta A, Jarrett M, Kadariya J, Xu H. Associations of Fecal Short Chain Fatty Acids With Colonic Transit, Fecal Bile Acid, and Food Intake in Irritable Bowel Syndrome. Clin Transl Gastroenterol. 2023 Jan 1;14(1):e00541. doi: 10.14309/ctg.0000000000000541. PMID 36227781